CLINICAL TRIAL: NCT05260385
Title: A Phase Ib / II Study to Evaluate the Efficacy and Safety of KC1036 in the Patients with Advanced Recurrent or Metastatic Digestive System Tumors
Brief Title: To Evaluate KC1036 in the Patients with Advanced Digestive System Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC1036-II-01
Record Dates: First submitted 2022-01-27; First posted 2022-03-02 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Digestive System Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QD regimen (Experimental): KC1036 was administered orally in 60 mg once daily, 21 days as a cycle.
  Interventions: Drug: KC1036
- BID regimen (Experimental): Dose-Escalation part : KC1036 was administered orally in 20 mg BID, 30 mg BID, or 40 mg BID.
  Dose-Expansion part : According to the results of Dose-Escalation, an appropriate BID regimen was selected for Dose-Expansion .
  Interventions: Drug: KC1036

INTERVENTIONS:
Drug: KC1036 — KC1036 are administered orally QD or BID in 21-day cycles.

SUMMARY:
The purpose of this study is to evaluate the preliminary efficacy, safety, tolerability and pharmacokinetics of KC1036 in participants with advanced recurrent or metastatic digestive system tumors.

DETAILED DESCRIPTION:
This is an open label, non-randomized，phase 1b/2 study to explore the preliminary antitumor activity of KC1036 in patients with advanced recurrent or metastatic digestive system tumors under BID or QD regimen.

The study will consist of two parts:

Part 1: QD regimen

To evaluate the efficacy and safety of KC1036 in the treatment of advanced recurrent, unresectable and / or metastatic digestive system tumors under 60mg QD regimen.

Part 2: BID regimen

Dose-Escalation part : To explore the safety of KC1036 under 20mg BID, 30mg BID and 40mg BID in patients with advanced recurrent or metastatic digestive system tumors.

Dose-Expansion part : According to the results of Dose-Escalation, an appropriate BID regimen was selected for Dose-Expansion to evaluate the effectiveness and safety of KC1036 in patients with advanced recurrent, unresectable and / or metastatic digestive system tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant digestive system tumors;
* Patients with advanced recurrent, unresectable and / or metastatic digestive system tumors who have failed standard or conventional treatment:( definition of treatment failure: intolerable toxic and side effects, disease progression during treatment recurrence after treatment);
* Eastern Cooperative Oncology Group performance status score of 0 or 1;
* Life expectancy > 12 weeks;
* BMI≥18.0;
* Has adequate Hematologic, renal, and hepatic function;
* Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* Any patient who is known to have central nervous system (CNS) metastasis with clinical symptoms;
* Other kinds of malignancies;
* Gastrointestinal abnormalitiest;
* Cardiovascular and cerebrovascular diseases;
* Previous treatment with small molecule vascular targeting inhibitor；
* Prior anti-tumor therapies with chemotherapy, radiotherapy, hormonotherapy, biotherapy, immunotherapy, operation within 4 weeks before enrollment;
* Involved in other clinical trials within 4 weeks before enrollment;
* Major surgical procedure, open biopsy, or significant traumatic injury 4 weeks before enrollment;
* Uncontrolled massive ascites,pleural/pericardial effusion;
* Uncontrolled ongoing or active bacterial, viral or fungal infectious; Fever of unknown cause (> 38.5 ℃) occurred within 2 weeks before enrollment;
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection ;
* Pregnant or lactating women or those who do not take contraceptives, including men;
* Any other metabolic dysfunction, abnormal physical examination findings, or clinical laboratory findings;
* Inability to comply with protocol required procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | approximately 2 year.
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | approximately 2 year
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | approximately 2 year.
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | approximately 2 year.
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.
Pharmacokinetics (PK) profile: Cmax | approximately 2 year.
  Parameters: Peak Plasma Concentration
Pharmacokinetics (PK) profile: Tmax | approximately 2 year.
  Parameters: Time to reach the maximum plasma concentration
Pharmacokinetics (PK) profile: T1/2 | approximately of 2 year.
  Parameters: Terminal half-life
Pharmacokinetics (PK) profile: AUC | approximately of 2 year.
  arameters: Area under the single-dose plasma concentration-time curve.
Adverse events (AEs) | approximately of 2 year.
  Incidence of treatment-related AEs

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - The first affiliated hospital of bengbu medical college, Bengbu
  - Chongqing University Three Gorges Hospital, Chongqing
  - Fujian Cancer Hospital, Fujian
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Henan
  - Hubei Cancer Hospital, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technologe, Hubei
  - Shandong Cancer Hospital & Institute, Shandong
  - Shanghai Chest Hospital, Shanghai
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen
  - Tianjin Medical University Cancer Institute &Hospital, Tianjin
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No